CLINICAL TRIAL: NCT05449028
Title: Helicobacter Pylori Eradication Therapy in Portugal: Prospective, Randomized, Blind and Multicentre Trial on the Efficacy of Quadruple Therapies and Their Clinical Impact, and Immunological and Gut Microbiota Changes
Brief Title: Helicobacter Pylori Eradication Therapy in Portugal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Principal Investigator, Elisa Gravito-Soares, Principal Investigator, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HpETIP
Record Dates: First submitted 2022-05-22; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Helicobacter Pylori; Gut Microbiota; Immunology
MeSH Terms: interventions — Bismuth

STUDY DESIGN:
Intervention Model Description: An interventional study is proposed to compare the efficacy and safety of the different approved H. pylori eradication quadruple regimens. Patients will be randomly assigned to the five quadruple regimens arms (A, B, C D and E). All patients will be followed during 12 months. A standardized protocol will be applied for all the groups, differing only in type of quadruple regimen used.
Who Masked: Participant, Investigator
Masking Description: Sampling: Consecutive sampling of incident cases of patients with H. pylori gastric infection and clinical indication for its eradication; Patients will be continuously monitored throughout the study. Regarding the evaluation of oral and gut microbiota and immunological changes, the study will be blinded, since the researchers responsible for sequencing and immunological analysis will not know the therapeutic scheme applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- H. pylori eradication scheme A (Experimental): Esomeprazole 40mg bid + amoxicillin 1g 12/12h + clarithromycin 500mg 12/12h + metronidazole 500mg 8/8h, for 14 days
  Interventions: Drug: H. pylori eradication scheme A
- H. pylori eradication scheme B (Experimental): Esomeprazole 40mg bid + amoxicillin 1g 12/12h + clarithromycin 500mg 12/12h + metronidazole 500mg 12/12h, for 14 days
  Interventions: Drug: H. pylori eradication scheme B
- H. pylori eradication scheme C (Experimental): Esomeprazole 40mg bid + bismuth subsalicylate 420mg 6/6h + metronidazole 375mg 6/6h + tetracycline 375mg 6/6h, for 10 days
  Interventions: Drug: H. pylori eradication scheme C
- H. pylori eradication scheme D (Experimental): Esomeprazole 40mg bid + amoxicillin 1g 12/12h for 7 days, followed by esomeprazole 40mg bid + clarithromycin 500mg 12/12h + metronidazole 500mg 12/12h for 7 days
  Interventions: Drug: H. pylori eradication scheme D
- H. pylori eradication scheme E (Experimental): Esomeprazole 40mg bid + amoxicillin 1g 12/12h for 7 days, followed by esomeprazole 40mg bid + amoxicillin 1g 12/12h + clarithromycin 500mg 12/12h + metronidazole 500mg 12/12h for 7 days
  Interventions: Drug: H. pylori eradication scheme E

INTERVENTIONS:
Drug: H. pylori eradication scheme A — Esomeprazole 40mg bid + amoxicillin 1g 12/12h + clarithromycin 500mg 12/12h + metronidazole 500mg 8/8h, for 14 days
  Other Names: Concomitant bismuth-free A
  Arms: H. pylori eradication scheme A
Drug: H. pylori eradication scheme B — Esomeprazole 40mg bid + amoxicillin 1g 12/12h + clarithromycin 500mg 12/12h + metronidazole 500mg 12/12h, for 14 days
  Other Names: Concomitant bismuth-free B
  Arms: H. pylori eradication scheme B
Drug: H. pylori eradication scheme C — Esomeprazole 40mg bid + bismuth subsalicylate 420mg 6/6h + metronidazole 375mg 6/6h + tetracycline 375mg 6/6h, for 10 days
  Other Names: Pylera; Concomitant with bismuth
  Arms: H. pylori eradication scheme C
Drug: H. pylori eradication scheme D — Esomeprazole 40mg bid + amoxicillin 1g 12/12h for 7 days, followed by esomeprazole 40mg bid + clarithromycin 500mg 12/12h + metronidazole 500mg 12/12h for 7 days
  Other Names: Sequential
  Arms: H. pylori eradication scheme D
Drug: H. pylori eradication scheme E — Esomeprazole 40mg bid + amoxicillin 1g 12/12h for 7 days, followed by esomeprazole 40mg bid + amoxicillin 1g 12/12h + clarithromycin 500mg 12/12h + metronidazole 500mg 12/12h for 7 days
  Other Names: Hybrid
  Arms: H. pylori eradication scheme E

SUMMARY:
Helicobacter pylori (H. pylori) infection remains a major public health problem, with an estimated prevalence of over 50% worldwide and 60-86% for Portugal. H. pylori is associated with significant morbidity and mortality from peptic ulcerative disease to gastric cancer, whose eradication therapy has proven to be effective in preventing these complications. Factors involved in the development of these conditions include H. pylori virulence, host genetic factors and gut microbiota. Given the increasing pattern of antibiotic resistance evidenced by this bacterium and the scarcity of available antibiotic therapy, both in Portugal and worldwide, there is not enough evidence on the best eradication strategy. Regarding the uncertainties about the potential negative impact of indiscriminate use of eradication therapy on gut microbiota, either by proton pump inhibitors or by antibiotics per se, there is an overriding need for evidence about the real impact of this therapy on oral or gut flora and possible clinical consequences in immunological, metabolic, nutritional and oncological terms.

Objectives: Comparative evaluation of the efficacy of the different quadruple therapy regimens recommended for the H. pylori eradication. Comparative evaluation of the safety profile in terms of clinical, and immunological and gut microbiota impact of the different therapies for the H. pylori eradication.

DETAILED DESCRIPTION:
Introduction: Helicobacter pylori (H. pylori) infection remains a major public health problem, with an estimated prevalence of over 50% worldwide and 60-86% for Portugal. H. pylori is associated with significant morbidity and mortality from peptic ulcerative disease to gastric cancer, whose eradication therapy has proven to be effective in preventing these complications. Factors involved in the development of these conditions include H. pylori virulence, host genetic factors and gut microbiota. Given the increasing pattern of antibiotic resistance evidenced by this bacterium and the scarcity of available antibiotic therapy, both in Portugal and worldwide, there is not enough evidence on the best eradication strategy. Regarding the uncertainties about the potential negative impact of indiscriminate use of eradication therapy on gut microbiota, either by proton pump inhibitors or by antibiotics per se, there is an overriding need for evidence about the real impact of this therapy on oral or gut flora and possible clinical consequences in immunological, metabolic, nutritional and oncological terms.

Objectives: Comparative evaluation of the efficacy of the different quadruple therapy regimens recommended for the H. pylori eradication. Comparative evaluation of the safety profile in terms of clinical, and immunological and gut microbiota impact of the different therapies for the H. pylori eradication.

Methods: Prospective longitudinal multicentre study of total of patients with gastric infection by H. pylori, diagnosed by 13C-urea breath test or histological analysis of gastric biopsies and clinical indication for its eradication, referred to the different participating Portuguese hospital units and a blind randomized controlled clinical trial of the efficacy and safety of the different quadruple therapy regimes recommended for the H. pylori eradication. This study will be carried out in 4 phases: Phase 1 - Recruitment and randomization of patients by the different quadruple eradication schemes with and without bismuth (5 parallel arms); Phase 2 - H. pylori eradication with evaluation of the efficacy and safety rates at 1 month and the absence of reinfection at 12 months after treatment and collection of stool samples before and after the eradication therapy for evaluation of changes in gut microbiota; Phase 3 - Analysis of richness, diversity and uniformity of gut microbiota by DNA sequencing using the hypervariable region of the ribosomal 16S bacteria gene as a taxonomic identification marker and their clinical impact on immunology, metabolism and nutrition at 12 months after the H. pylori eradication therapy; and Phase 4 - Analysis of immunological changes through the study of cell populations by flow cytometry (CD4+, CD8+, B-cell, T-cell, natural killer cells, cells ratio) and cytokines, chemokines and growth factors by xMAP/Luminex before and 12 months after the H. pylori eradication therapy.

Expected results, impact and scientific outputs: Given the high rate of triple therapy inefficacy, high antibiotic resistance and the scarcity and controversy of existing literature on quadruple regimens, there may be relevant differences in the approved quadruple regimens for the H. pylori eradication, being necessary to define which is the most effective and safe in Portugal, decreasing the rate of ineffectiveness and exposure to multiple antibiotics. The homeostasis of gut microbiota is significantly changed after H. pylori eradication and this modification may be substantially different according to the therapeutic scheme used, with clinical implications on immunology, metabolism and nutrition. Thus, a randomized trial to compare quadruple regimens is need, allowing in the future, an individualized selection of the H. pylori eradication regimen, taking into account the higher efficacy and safety and lower gut dysbiosis and its systemic consequences, in short and long term. Modulating oral and gut microbiota therapies, including prebiotics, probiotics, symbiotics, fecal microbiota transplantation and perhaps targeted-immunotherapy may be beneficial as adjuvant therapy to existing H. pylori eradication regimens, in a systematic way or for some therapeutic regimes or risk groups.

ELIGIBILITY:
Inclusion Criteria:

* Gastric infection by H. pylori by histological examination of gastric biopsies or carbon 13-labeled urea breath test.

Exclusion Criteria:

* Age < 18 years;
* Pregnant, breast-feeding or women of childbearing age who do not comply with effective anticonception measures;
* History of allergy, hypersensitivity or contraindication to the use of H. pylori eradication drugs (antibiotics or proton pump inhibitors);
* History of previous gastrointestinal surgery or neoplasia;
* Previous H. pylori eradication therapies; Antibiotic or probiotic therapies in the month prior to recruitment;
* Use of proton pump inhibitors, other antacids or gastric mucosal protection agents in the 2 weeks prior to recruitment;
* Corticosteroids or immunomodulatory therapy in the month prior to recruitment;
* Immunodeficiency;
* Insulin-treated diabetes mellitus;
* Obesity (Body mass index ≥30Kg/m2);
* Use of laxative therapy in the 15 days prior to recruitment;
* Decompensated heart, liver, kidney or respiratory diseases and;
* Refusal or inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy assessed by the eradication rate of the different therapeutic regimens recommended as H. pylori eradication therapy | 1 month after the intervention
  Efficacy rate of H. pylori eradication will be determined for five different therapeutic regimens (sequential, hybrid and concomitants with or without bismuth). A successful eradication implies no documentation of H. pylori by carbon 13-labeled urea breath test or upper gastrointestinal endoscopy with biopsies, depending on clinical indication, at 1 month after H. pylori eradication (D40 or D44). A therapeutic regimen will be considered effective if it achieves more than 90% of H. pylori eradication (the minimum efficacy rate).
Efficacy assessed by the re-infection rate after the different therapeutic regimens recommended as H. pylori eradication therapy | 12 months after the intervention
  At 12 months after H. pylori eradication, a carbon 13-labeled urea breath test will be performed to exclude re-infection.
Safety assessed by overall treatment-adverse events and and severe treatment-adverse events rates of the different therapeutic regimens recommended as H. pylori eradication therapy | 1 month after the intervention
  Safety profile of H. pylori eradication will be determined for five different therapeutic regimens measuring adverse effects according to Medical Dictionary for Regulatory Activities (MedDRa). Therapy-related adverse events and its severity (by visual analogue scale of intolerance [0-10] and classification of the severity of adverse effects for the daily life activities according to [BoThBo96]) will be recorded at 1 month post-eradication follow-up.
Safety assessed by overall treatment completion rate of the different therapeutic regimens recommended as H. pylori eradication therapy | 1 month after the intervention
  Safety profile of H. pylori eradication will be determined for five different therapeutic regimens measuring the treatment completion rate to the treatment at 1 month post-eradication follow-up.

SECONDARY OUTCOMES:
Post-eradication changes assessed by OTU and their relative abundance in gut microbiota | Changes from baseline at immediately after the intervention
  Stool samples shall be collected, stored at -20°C and then analyzed on 3 occasions: 1) baseline, 2) after stopping treatment (D10 or 14) and 3) 1 month after treatment (D40 or 44). A standard protocol with the conditions of collection, storage and transport of the different collected samples will be used. Analysis of gut microbiota by DNA sequencing using the hypervariable region of the 16S ribosomal bacteria gene as a taxonomic identification marker by bioinformatic analysis, for taxonomic identification and determination of the relative abundance of each Operational Taxonomy Units (OTU). The gut microbiota will be evaluated by an independent operator who does not know the therapeutic scheme used.
Post-eradication changes assessed by OTU and their relative abundance in gut microbiota | Changes from baseline at 1 month after the intervention
  Stool samples shall be collected, stored at -20°C and then analyzed on 3 occasions: 1) baseline, 2) after stopping treatment (D10 or 14) and 3) 1 month after treatment (D40 or 44). A standard protocol with the conditions of collection, storage and transport of the different collected samples will be used. Analysis of gut microbiota by DNA sequencing using the hypervariable region of the 16S ribosomal bacteria gene as a taxonomic identification marker by bioinformatic analysis, for taxonomic identification and determination of the relative abundance of each Operational Taxonomy Units (OTU). The gut microbiota will be evaluated by an independent operator who does not know the therapeutic scheme used.

OTHER OUTCOMES:
Post-eradication changes assessed by immunological cells populations in immunological profile | Changes from baseline at 12 months after the intervention
  Fresh peripheral blood samples will be collected and analyzed on 2 occasions: 1) baseline and 2) 12 months after treatment. A standard protocol with the conditions of collection, storage and transport of the different collected samples will be used. Analysis of immunological changes: Immunological profile will be analysed through the study of cell populations (CD4+, CD8+, B-cell, T-cell, natural killer cells, cells ratio) by multiparametric flow cytometry, before and 12 months after the H. pylori eradication therapy, by an independent operator who does not know the therapeutic scheme used.
Post-eradication changes assessed by cytokines, chemokines and growth factors in immunological profile | Changes from baseline at 12 months after the intervention
  Fresh peripheral blood samples will be collected and analyzed on 2 occasions: 1) baseline and 2) 12 months after treatment. A standard protocol with the conditions of collection, storage and transport of the different collected samples will be used. Analysis of immunological changes: Immunological profile will be analysed through the study of cytokines, chemokines and growth factors by xMAP/Luminex, before and 12 months after the H. pylori eradication therapy, by an independent operator who does not know the therapeutic scheme used.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Gravito-Soares, MD, Principal Investigator — Unidade Local de Saúde de Coimbra, EPE
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
No applicable.

REFERENCES:
- [Result] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Result] Zamani M, Ebrahimtabar F, Zamani V, Miller WH, Alizadeh-Navaei R, Shokri-Shirvani J, Derakhshan MH. Systematic review with meta-analysis: the worldwide prevalence of Helicobacter pylori infection. Aliment Pharmacol Ther. 2018 Apr;47(7):868-876. doi: 10.1111/apt.14561. Epub 2018 Feb 12. PMID 29430669
- [Result] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Result] Gao JJ, Zhang Y, Gerhard M, Mejias-Luque R, Zhang L, Vieth M, Ma JL, Bajbouj M, Suchanek S, Liu WD, Ulm K, Quante M, Li ZX, Zhou T, Schmid R, Classen M, Li WQ, You WC, Pan KF. Association Between Gut Microbiota and Helicobacter pylori-Related Gastric Lesions in a High-Risk Population of Gastric Cancer. Front Cell Infect Microbiol. 2018 Jun 19;8:202. doi: 10.3389/fcimb.2018.00202. eCollection 2018. PMID 29971220
- [Result] Chey WD, Leontiadis GI, Howden CW, Moss SF. ACG Clinical Guideline: Treatment of Helicobacter pylori Infection. Am J Gastroenterol. 2017 Feb;112(2):212-239. doi: 10.1038/ajg.2016.563. Epub 2017 Jan 10. PMID 28071659
- [Result] Savoldi A, Carrara E, Graham DY, Conti M, Tacconelli E. Prevalence of Antibiotic Resistance in Helicobacter pylori: A Systematic Review and Meta-analysis in World Health Organization Regions. Gastroenterology. 2018 Nov;155(5):1372-1382.e17. doi: 10.1053/j.gastro.2018.07.007. Epub 2018 Jul 7. PMID 29990487
- [Result] Lopo I, Libanio D, Pita I, Dinis-Ribeiro M, Pimentel-Nunes P. Helicobacter pylori antibiotic resistance in Portugal: Systematic review and meta-analysis. Helicobacter. 2018 Aug;23(4):e12493. doi: 10.1111/hel.12493. Epub 2018 Jun 17. PMID 29911329
- [Result] Almeida N, Romaozinho JM, Donato MM, Luxo C, Cardoso O, Cipriano MA, Marinho C, Fernandes A, Calhau C, Sofia C. Helicobacter pylori antimicrobial resistance rates in the central region of Portugal. Clin Microbiol Infect. 2014 Nov;20(11):1127-33. doi: 10.1111/1469-0691.12701. Epub 2014 Jul 12. PMID 24890952
- [Result] Graham DY, Lee YC, Wu MS. Rational Helicobacter pylori therapy: evidence-based medicine rather than medicine-based evidence. Clin Gastroenterol Hepatol. 2014 Feb;12(2):177-86.e3; Discussion e12-3. doi: 10.1016/j.cgh.2013.05.028. Epub 2013 Jun 8. PMID 23751282
- [Result] Cerqueira RM, Manso MC, Correia MR, Fernandes CD, Vilar H, Nora M, Martins P. Helicobacter pylori eradication therapy in obese patients undergoing gastric bypass surgery--fourteen days superior to seven days? Obes Surg. 2011 Sep;21(9):1377-81. doi: 10.1007/s11695-010-0254-4. PMID 20838918
- [Result] Almeida N, Donato MM, Romaozinho JM, Luxo C, Cardoso O, Cipriano MA, Marinho C, Fernandes A, Calhau C, Sofia C. Beyond Maastricht IV: are standard empiric triple therapies for Helicobacter pylori still useful in a South-European country? BMC Gastroenterol. 2015 Feb 15;15:23. doi: 10.1186/s12876-015-0245-y. PMID 25886722
- [Result] Boal Carvalho P, Magalhaes J, Dias de Castro F, Rosa B, Cotter J. Randomized Controlled Trial for Helicobacter pylori Eradication in a Naive Portuguese Population: Is Sequential Treatment Superior to Triple Therapy in Real World Clinical Setting? Acta Med Port. 2017 Mar 31;30(3):185-189. doi: 10.20344/amp.8072. Epub 2017 Mar 31. PMID 28550827
- [Result] Cerqueira RM, Correia M, Vilar H, Manso MC. Cumulative Helicobacter Pylori Eradication Rates by Adopting First- and Second- Line Regimens Proposed by the Maastricht IV Consensus in Obese Patients Undergoing Gastric Bypass Surgery. Obes Surg. 2018 Mar;28(3):743-747. doi: 10.1007/s11695-017-2915-z. PMID 29076008
- [Result] Heimesaat MM, Fischer A, Plickert R, Wiedemann T, Loddenkemper C, Gobel UB, Bereswill S, Rieder G. Helicobacter pylori induced gastric immunopathology is associated with distinct microbiota changes in the large intestines of long-term infected Mongolian gerbils. PLoS One. 2014 Jun 18;9(6):e100362. doi: 10.1371/journal.pone.0100362. eCollection 2014. PMID 24941045
- [Result] Myllyluoma E, Ahlroos T, Veijola L, Rautelin H, Tynkkynen S, Korpela R. Effects of anti-Helicobacter pylori treatment and probiotic supplementation on intestinal microbiota. Int J Antimicrob Agents. 2007 Jan;29(1):66-72. doi: 10.1016/j.ijantimicag.2006.08.034. Epub 2006 Dec 1. PMID 17141481
- [Result] Yap TW, Gan HM, Lee YP, Leow AH, Azmi AN, Francois F, Perez-Perez GI, Loke MF, Goh KL, Vadivelu J. Helicobacter pylori Eradication Causes Perturbation of the Human Gut Microbiome in Young Adults. PLoS One. 2016 Mar 18;11(3):e0151893. doi: 10.1371/journal.pone.0151893. eCollection 2016. PMID 26991500
- [Result] Hojo M, Asahara T, Nagahara A, Takeda T, Matsumoto K, Ueyama H, Matsumoto K, Asaoka D, Takahashi T, Nomoto K, Yamashiro Y, Watanabe S. Gut Microbiota Composition Before and After Use of Proton Pump Inhibitors. Dig Dis Sci. 2018 Nov;63(11):2940-2949. doi: 10.1007/s10620-018-5122-4. Epub 2018 May 24. PMID 29796911
- [Result] Buzas GM. Metabolic consequences of Helicobacter pylori infection and eradication. World J Gastroenterol. 2014 May 14;20(18):5226-34. doi: 10.3748/wjg.v20.i18.5226. PMID 24833852
- [Result] Chen L, Xu W, Lee A, He J, Huang B, Zheng W, Su T, Lai S, Long Y, Chu H, Chen Y, Wang L, Wang K, Si J, Chen S. The impact of Helicobacter pylori infection, eradication therapy and probiotic supplementation on gut microenvironment homeostasis: An open-label, randomized clinical trial. EBioMedicine. 2018 Sep;35:87-96. doi: 10.1016/j.ebiom.2018.08.028. Epub 2018 Aug 23. PMID 30145102
- [Result] Jakobsson HE, Jernberg C, Andersson AF, Sjolund-Karlsson M, Jansson JK, Engstrand L. Short-term antibiotic treatment has differing long-term impacts on the human throat and gut microbiome. PLoS One. 2010 Mar 24;5(3):e9836. doi: 10.1371/journal.pone.0009836. PMID 20352091
- [Result] Wang AY, Peura DA. The prevalence and incidence of Helicobacter pylori-associated peptic ulcer disease and upper gastrointestinal bleeding throughout the world. Gastrointest Endosc Clin N Am. 2011 Oct;21(4):613-35. doi: 10.1016/j.giec.2011.07.011. PMID 21944414
- [Result] Satoh Y, Ogawara H, Kawamura O, Kusano M, Murakami H. Clinical Significance of Peripheral Blood T Lymphocyte Subsets in Helicobacter pylori-Infected Patients. Gastroenterol Res Pract. 2012;2012:819842. doi: 10.1155/2012/819842. Epub 2012 Mar 28. PMID 22536220
- [Result] Carbo A, Bassaganya-Riera J, Pedragosa M, Viladomiu M, Marathe M, Eubank S, Wendelsdorf K, Bisset K, Hoops S, Deng X, Alam M, Kronsteiner B, Mei Y, Hontecillas R. Predictive computational modeling of the mucosal immune responses during Helicobacter pylori infection. PLoS One. 2013 Sep 5;8(9):e73365. doi: 10.1371/journal.pone.0073365. eCollection 2013. PMID 24039925
- [Result] Bagheri N, Salimzadeh L, Shirzad H. The role of T helper 1-cell response in Helicobacter pylori-infection. Microb Pathog. 2018 Oct;123:1-8. doi: 10.1016/j.micpath.2018.06.033. Epub 2018 Jun 21. PMID 29936093
- [Result] Song M, Rabkin CS, Torres J, Kemp TJ, Zabaleta J, Pinto LA, Hildesheim A, Sanchez-Figueroa L, Guarner J, Herrera-Goepfert R, Parsonnet J, Camargo MC. Circulating inflammation-related markers and advanced gastric premalignant lesions. J Gastroenterol Hepatol. 2019 May;34(5):852-856. doi: 10.1111/jgh.14518. Epub 2018 Nov 18. PMID 30357905
- [Result] Jafarzadeh A, Larussa T, Nemati M, Jalapour S. T cell subsets play an important role in the determination of the clinical outcome of Helicobacter pylori infection. Microb Pathog. 2018 Mar;116:227-236. doi: 10.1016/j.micpath.2018.01.040. Epub 2018 Jan 31. PMID 29407232
- [Result] Goll R, Cui G, Olsen T, Isaksen V, Gruber F, Husebekk A, Florholmen J. Alterations in antral cytokine gene expression in peptic ulcer patients during ulcer healing and after Helicobacter pylori eradication. Scand J Immunol. 2008 Jan;67(1):57-62. doi: 10.1111/j.1365-3083.2007.02037.x. Epub 2007 Nov 20. PMID 18028289
- [Result] de Boer WA, Thys JC, Borody TJ, Graham DY, O'Morain C, Tytgat GN. Proposal for use of a standard side effect scoring system in studies exploring Helicobacter pylori treatment regimens. Eur J Gastroenterol Hepatol. 1996 Jul;8(7):641-3. PMID 8853251

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT05449028/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT05449028/ICF_001.pdf